CLINICAL TRIAL: NCT05263011
Title: Effects of an Evening Snack Containing Avocado on Risk Factors for Diabetes in a Prediabetic Population
Brief Title: Avocado Snacks in a Prediabetic Population
Acronym: AVOC4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Hass Avocado Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB-2021-81
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: PreDiabetes
Keywords: avocado
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Avocado snack (Experimental): 1 avocado
  Interventions: Other: Avocado
- control snack + fiber supplement + vegetable oil (Placebo Comparator): high fat, high fiber control
  Interventions: Other: low fat yogurt + fiber +fat
- control snack (Other): Low-fiber, low-fat
  Interventions: Other: low fat yogurt

INTERVENTIONS:
Other: Avocado — 1 avocado as evening snack
  Arms: Avocado snack
Other: low fat yogurt — 1 serving of low fat yogurt matching calories of 1 avocado
  Arms: control snack
Other: low fat yogurt + fiber +fat — low fat yogurt mixed with ultra processed olive oil + fiber supplement, equivalent to fat and fiber content in 1 avocado
  Arms: control snack + fiber supplement + vegetable oil

SUMMARY:
Compare the effects of three evening snacks on morning fasting and postprandial glucose and insulin concentrations in individuals with prediabetes.

DETAILED DESCRIPTION:
The study is a single-center, randomized, single-blinded, 3-arm, and cross-over study design. Participants will be randomized to receive three eventing snack in randomized order: low-fiber, low-fat control snack (low-fat yogurt); whole avocado snack; or control snack + fiber supplement + vegetable oil, which will be consumed in the evening before the clinic visit. Twelve hours (12 h) after snack intake (based on subjects typical evening snack and morning breakfast routine), participants will report to the clinic for fasting blood draws, followed by a standard meal with a minimum of 50 g available carbohydrate, and repeated blood collection for 3 hours. On the day of "snack" intervention (ie., 24 h before standard meal testing), subjects will be guided to follow their typical dietary pattern in consultation with staff. Food diaries with a general plan will be used as a tool to help with dietary compliance.

STUDY PROCEDURES: SCREENING VISIT:

Interested subjects will be asked to come to the Clinical Nutrition Research Center (CNRC) on the IIT Campus, Chicago, IL, where the study will take place for a screening visit to determine if they are eligible to participate in the study. The screening visit will take 2 hours. Prospective subjects must read, sign and date a written Institutional Review Board (IRB) approved Informed Consent Form prior to performing any study procedure.

At the on-site screening visit, subject will be asked to arrive after overnight fasting for 10-12 hours and be well-hydrated. Subject will be instructed to aim for a water intake of at least 8-10 cups for the 24 hours before the screening visit. Determining eligibility to participate includes having subjects to complete a series of questionnaires related to their health, medication use, dietary habits, and physical activity history. Anthropometrics (height, weight and waist circumference), body composition, ear temperature, and vital signs (blood pressure and heart rate) will be measured. For women under the age of 60 years, a pregnancy test will be conducted. Body mass index (BMI) will be calculated from height and weight measurements. Fasting blood glucose level by capillary blood from finger prick will be tested. For vital sign measurements, subjects will sit in a comfortable chair, feet uncrossed and on the floor and will be asked to rest quietly for 5 minutes before measuring blood pressure and heart rate. Arm vein will be assessed using a vein access scale test. Subject will be instructed to complete a 24-hour food recall.

Based on the results of the questionnaires, BMI calculation, and health evaluation, subjects who meet the inclusion and exclusion criteria will be invited to participate in the study. Eligible subjects will be trained and instructed to record all food and beverages consumed for a 24 hour period on food record diarie using ASA24. Subjects will be asked not to take any allergy medications and/or any pain medications such as Aspirin, Excedrin, Ibuprofen (Advil, Motrin, Nuprin), Naproxen, or Aleve within 48 hours of each scheduled study days. Tylenol is allowed. If they need to take allergy/pain medication 48 hours prior to their study day, we will ask them to let the study investigators know so they can be rescheduled. Before leaving the CNRC, subjects will be provided with written instruction for "how to prepare for your study visit". This will include instructions for eating a standardized dinner meal the night before the study day, consume the assigned study snacks, fasting overnight (10-12 hours), avoidance of vigorous physical activity, alcoholic and caffeinated beverage consumption for at least 24 hours preceding a study day, maintain regular sleep pattern and usual diet except for the guidance provided for "foods and beverages to avoid or limit". If subject did not get enough sleep during the night preceding a study day, we will ask them to let us know so we can reschedule their study day.

STUDY DAYS:

Participation in this study will last approximately 2 to 3 weeks and include 3 Study Day visits to the CNRC. Each Study Day visit will last about ~3.5 hours.

The day before each of the Study Day visits, subjects will be asked to come to the Center to pick up a dinner meal and evening snack and will be asked to consume only the provided dinner meal and snacks the evening before the visit. Subject will be provided with guidance on how to maintain the same dinner intake, and when to consume the snacks (12 hour before the scheduled study visit time, schedule based on the subject's typical evening snack and morning breakfast routine) At each Study Day visit, subjects will arrive at the clinic after fasting for 10 to 12 hours and in a well-hydrated and well-rested state after regular sleep the night before. If they are taking medication(s) each morning, they will be asked not to take the medication(s) at home and instead to bring to the CNRC to be taken in the presence of the study investigator so the medications(s) is taken at the same time before each Study Day visit.

Study protocol adherence will be corroborated by asking about the period of fasted state. Subject will also be asked about their detailed food intake the 24-hour period prior to the visit to ensure consistency and compliance with the protocol requirements. Subjects experiencing unusual stressful events (such as loss of job, loss of loved one, divorce, etc...) or having active infection will be rescheduled to a later time agreed upon by the subject and investigator. Participants having experienced active infection can be rescheduled when symptoms have been gone for at least 5 days and been off treatment (ex. Antibiotics) for same time duration. The test period will be extended for study completion in these cases. Subject will be asked about their medication intake and health status since their last visit to ensure that subjects are maintaining their good health and medication intake.

After confirming compliance with the protocol, anthropometric measurements, and vital signs (blood pressure, heart rate and ear temperature) will be taken. A finge prick for fasting blood glucose will be taken to confirm if the subject is fasting. A licensed healthcare professional (LHCP) will evaluate and place a catheter on the antecubital site of the subject's non-dominant arm or arm of preference by subject. A catheter is a thin flexible tube that allows sampling of blood through one port throughout the Study Day. Once the catheter is placed, a blood sample will be taken (Time point T 0). After completing baseline blood sampling, subjects will receive a standard meal with a minimum of 50 g available carbohydrate to consume within 10 minutes. After the test food is consumed, additional blood samples will be taken at 15, 30, 45, 60, 90, 120, 180 minutes after the start of breakfast consumption. Subjects are allowed to drink water and the amount will be recorded. After completion of all study procedures and data/sample collection for the day, the catheter will be removed and subjects will be evaluated for safety and/or discomfort/symptoms before leaving the study site. They will be given a snack and written instructions in preparation for the next visit. Study day visits will be scheduled at least 3 days apart. Study Day 2 and 3 will be exactly the same as Study Day 1 except the evening snacks to consume before each Study Day. Blood collection: Blood will be collected a total of 7 times on each Study Day visit and 4 mL of the blood sample will be collected at each time point at each Study Day visit. Over the course of the whole study, the total amount of blood collected will be ~84 mL, which is less than what is allowed for a one-time blood donation (~550 mL).

Adverse Events (AEs) will be assessed throughout Study Day visit. In an emergency while the study subject is at CNRC, a LHCP will be on site to monitor the subject. In the unlikely event of a medical emergency, 911 and emergency response will be called to the site. The adverse event will be documented, determined as treatment-related or non-treatment related by the Investigator and submitted to the IRB within 3 days or sooner for treatment related adverse events. Serious adverse events (SAE) will be reported within 24 hours of our knowledge of the SAE. A copy will be filed in the subject's study chart. Study staffs are also trained and certified in CPR techniques.

In the event of an after-hours emergency, subject will be advised to obtain medical attention as appropriate for the described symptoms. The subject is not required to contact the Investigator prior to seeking medical attention, however will be required to report the adverse event to the study manager or study coordinator at the next scheduled contact or sooner if appropriate.

Retention and Compliance:

This study will include periodic telephone reminder calls along with in-person contact for study day visits. Phone calls will be made to remind subjects to record food intake (according to the subject specific pre-determined food record schedule), maintain consistency in their overall diet and exercise habit prior to the Study Day visit and to confirm visit schedules.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 25-70 years
* Fasting blood glucose concentration between 100 mg/dL and 125 mg/dL at screening visit
* Blood pressure 120-160 mmHg systolic or 80-100 mm/Hg diastolic at screening visit
* Nonsmokers (past smokers can be allowed if they have abstinence for minimum of 12 months)
* Judged to be in good health on the basis of the medical history (i.e., no clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease)
* Not taking any medications that would interfere with outcomes of the study, (e.g., lipid lowering medications, anti-inflammatory drugs, dietary supplements, etc.)
* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol (follow the dietary plans, come to scheduled visits, record food intake in a diary, complete questionnaires, provide blood samples and complete other tests (eye and brain/cognitive function)
* Able to maintain usual physical activity pattern
* Able to abstain from alcohol consumption and avoid vigorous physical activity for 24 hours prior to and during the study visit

Exclusion Criteria:

* Men and women who have blood pressure >160 mmHg (systolic)/100 mmHg (diastolic) at screening visit
* Men and women who have fasting blood glucose concentration <100 or >125 mg/dL at screening visit
* Men and women with diabetes
* History of a cardiovascular event, respiratory, renal, gastrointestinal, hepatic or eye disease or surgery (e.g., heart failure, myocardial infarction, stroke, angina, related surgeries, etc.) that, in the opinion of the investigator, could interfere with the interpretation of the study results
* Head injury in past 6 months
* Men and women with cancer other than non-melanoma skin cancer in previous 5 years
* Taking medication or dietary supplements that may interfere with the outcomes of the study, (e.g., antioxidant supplement, anti-inflammation, lipid-lowering medication, blood pressure-lowering medication, etc.). Subjects may choose to go off dietary supplements (requires 30-day washout; e.g., fish oil, etc.)
* Vegan or other extreme dietary regimens (e.g., Atkins diet, etc.) as judged by the investigator
* Known or suspected intolerance, allergies or hypersensitivity to study foods or treatments
* Current smoker or smoked/vaped within the last 12 months
* Unstable weight: Actively losing or gaining weight or trying to lose or gain weight. Gained or lost weight +/- 5 kg (11 lbs.) in previous 2 months.
* Substance (alcohol or drug) abuse within the last 2 years
* Present with significant psychiatric or neurological disturbances
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are lactating
* Major trauma or a surgical event within 2 months or longer depending on trauma or event and after consultation with PI.
* Has used antibiotics within the previous 2 months
* History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional
* Excessive coffee and tea consumers (> 4 cups/d)
* Donated blood within last 3 months
* Men and women who do excessive exercise regularly or are an athlete
* Women who are taking unstable dose and brand of hormonal contraceptives and/or stable dose and brand less than 6 months
* Unusual working hours (e.g., working overnight; 3rd shift)

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Changes in plasma glucose concentration | time 0-180 minutes
  will be analyzed by a Randox automated clinical analyzer
Changes in plasma insulin concentration | time 0-180 minutes
  will be analyzed by a Randox automated clinical analyzer
Changes in plasma triglycerides concentration | time 0-180 minutes
  will be analyzed by a Randox automated clinical analyzer
Changes in plasma Interleukin (IL)-6 concentration | time 0-3 hours
  will be analyzed by ELISA or EIA using purchased kits and reagents from R&D systems
Changes in plasma tumor necrosis factor (TNF)-alpha, concentration | time 0-3 hours
  will be analyzed by ELISA or EIA using purchased kits and reagents from R&D systems

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Preiss C, Marquis O, Edirisinghe I, Burton-Freeman BM. Using the Avocado as an Evening Snack to Investigate Whole Food Matrix and Macronutrient Composition on Morning Metabolic Indices in Adults With Prediabetes. Curr Dev Nutr. 2025 Jun 12;9(7):107486. doi: 10.1016/j.cdnut.2025.107486. eCollection 2025 Jul. PMID 40689342